CLINICAL TRIAL: NCT06540625
Title: Validation of a Novel Handheld Device for Accurate Cricoid Pressure in Healthy Volunteers
Status: Not yet recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 4991
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cricoid Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: the use of CP device application on human subjects. — Trained providers will be asked to apply CP at 10N of force to the marked location using the cricoid applicator for one minute. Data relating to applied force across the whole one minute will be measured continuously and will be captured and stored. The CP device will have a microdisc port for internal memory and then the wifi on the board will transfer the information to a cloud server for backup and storage for redundancy.
  A threshold of 10 ± 2 N applied force will be set to define successful CP attempts. Participants must remain in this range for 95% of the trial time after the first five seconds have passed.
  At any point during the CP application, if the volunteer experiences pain, they can request that the pressure be stopped. However, we do not expect any pain with 10N, except for minor discomfort.

SUMMARY:
Pulmonary aspiration of gastric contents is a leading cause of anesthesia-related morbidity and mortality, particularly in emergency surgeries and among patients who are not appropriately fasted prior to airway intervention. The application of cricoid pressure (CP), also known as the "Sellick maneuver" is the current clinical practice to prevent aspiration of gastric content during Rapid-sequence induction (RSI) of general anesthesia. This conventional CP uses manual pressure over the cricoid cartilage during RSI procedure for patients at high risk of aspiration. Since its incorporation into clinical practice, the utility and technique of CP have garnered considerable debate, mainly due to the inability to standardize the magnitude and consistency of the applied force. Too little force may be ineffective at preventing regurgitation and excessive force may impede ventilation and actually worsen laryngoscopy views, making intubation more difficult.

A significant challenge in current clinical practice of CP is the inconsistency in the force applied, which often falls short of the necessary intensity and duration. To address this issue, we developed a groundbreaking handheld device capable of monitoring applied pressure in real-time, aiding providers in delivering precise and reproducible CP. Furthermore, our device utilizes sensor fabrication technology, integrating microelectronic systems and microprocessors to measure and display force in real-time, all while remaining portable. However, before implementation in clinical practice, rigorous testing through human volunteer studies and subsequent clinical trials is imperative. Hence, this study aims to validate the efficacy of our novel CP device in helping Providers apply the accurate target force.

DETAILED DESCRIPTION:
The investigators have developed a clinically robust, customizable, handheld device that incorporates a micro load cell (a sensor to measure force) and Arduino processor (a small circuit board) in order to apply accurate and reproducible CP. The novel device contains a compression/tension micro load cell (model: TAS520-5kg HT Sensor Technology Co. Ltd.) that is incorporated into a 3D printed CP application system (Figure 1). The 3D printed cricoid neck pad is designed based on average cricoid cartilage dimensions.16 The device is designed for testing forces in the range of 0-5 kg (~50 N). The load cell system is then attached to an Arduino circuit board, HX711 load cell amplification circuit and LCD digital display that are all encased in a 3D printed enclosure. The device has a microdisc port for internal memory that allows transfer of data for further backup and analysis. The device uses a rechargeable battery for ease of use and portability. The Force (N) is displayed on the LCD screen to give the user the exact force being applied in real time.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia department staff Volunteers Participants
* Perioperative staff Volunteers Providers

Exclusion Criteria:

* Participants with skin problems, such as eczema or psoriasis
* Participants who is pregnant
* Participants with a history of neck or throat injury or anatomical abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Participants Participants will include staff volunteers from the Department of Anesthesia at two participating hospitals. A recruitment email will be distributed by the site study Research Coordinator to the department staff including research staff, administrative staff, anesthesia staff, anesthesia assistants, fellows, residents, and nurses.
  * Providers Providers will include volunteers from perioperative staff consisting of operating room nurses, anesthesia staff, anesthesia assistants, fellows and residents who perform CP during RSI at the participating hospital. Perioperative staff who have previously applied CP or received training in CP will be included in this study.
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess whether the Providers can use the CP device with an accurate target force and maintain the force in an acceptable range over one minute. | one day
  We set a target of 10N force for the study, with an acceptable range of 10N ± 2N.

SECONDARY OUTCOMES:
Usability of the device based on feedback from both Participants and Providers | one day
  Proportion of Providers who think CP device will be useful in clinical practice
Effectiveness of the video training based on feedback from Providers | One day
  Proportion of Providers who think the video training was useful

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dinsmore, MD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No